CLINICAL TRIAL: NCT04613518
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Efficacy, and Biomarker Response of BMS-986165 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: A Study of the Safety, Efficacy, and Biomarker Response of BMS-986165 in Participants With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-127; 2019-004878-26 (EudraCT Number); U1111-1245-2970 (Other: World Health Organization)
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator
- Open label Extension, BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Specified Dose on Specified Days
  Arms: BMS-986165; Open label Extension, BMS-986165
Other: Placebo Comparator — Specified Dose on Specified Days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability, efficacy, and biomarker response of BMS-986165 administered orally in participants with moderate to severe ulcerative colitis. The study was originally designed to test deucravacitinib at two doses for 12 weeks compared to placebo. After the initial 12-Week period, all subjects receive active therapy (open-label extension). With protocol amendment 2, one of the dose treatment arms is being removed from the 12-week double blind period with no change to the open-label extension.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ulcerative colitis (UC) at least 3 months' duration prior to screening
* Moderately to severely active UC as assessed by the modified Mayo score
* Documentation of an inadequate response, loss of response, or intolerance to a treatment course of 1 or more of the following standard of care medications: oral 5-aminosalicylic acids, corticosteroids, immunomodulators, anti-tumor necrosis factor (TNF) agents, integrin inhibitors[SA1]
* Documentation of prior treatment with corticosteroids for ≥ 4 weeks
* Males and females must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Current diagnosis of Crohn's disease (CD) or diagnosis of indeterminate colitis (IC), ischemic colitis, or pseudomembranous colitis
* Current evidence of fulminant colitis, abdominal abscess, toxic megacolon, or bowel perforation
* History or evidence of any extensive colonic resection, or subtotal or total colectomy
* Women who are pregnant or breastfeeding
* Prior exposure to BMS-986165 or a tyrosine kinase 2 (TYK2) inhibitor

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (26):
- United States (10):
  - Local Institution - 0014, San Diego, California
  - Local Institution - 0036, Arlington Heights, Illinois
  - Local Institution - 0016, Shreveport, Louisiana
  - Local Institution - 0015, New York, New York
  - Local Institution - 0026, Chapel Hill, North Carolina
  - Local Institution - 0013, Cleveland, Ohio
  - Local Institution - 0020, Oklahoma City, Oklahoma
  - Local Institution - 0032, Garland, Texas
  - Local Institution - 0039, Lubbock, Texas
  - Local Institution - 0033, Southlake, Texas
- Australia (2):
  - Local Institution - 0005, Sydney, New South Wales
  - Local Institution - 0002, Camberwell, Victoria
- Canada (3):
  - Local Institution - 0007, Edmonton, Alberta
  - Local Institution - 0025, London, Ontario
  - Local Institution - 0008, Vaughan, Ontario
- Germany (3):
  - Local Institution - 0003, Berlin
  - Local Institution - 0019, Dresden
  - Local Institution - 0006, Kiel
- Local Institution - 0009, Amsterdam, North Holland, Netherlands
- Poland (4):
  - Local Institution - 0031, Warsaw, Masovian Voivodeship
  - Local Institution - 0030, Warsaw, Masovian Voivodeship
  - Local Institution - 0029, Bydgoszcz
  - Local Institution - 0028, Bydgoszcz
- Local Institution - 0011, San Juan, Puerto Rico
- United Kingdom (2):
  - Local Institution - 0023, London, England
  - Local Institution - 0027, Cambridge

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04613518.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: BMS-986165 6 mg BID arm was removed under Protocol Amendment 02.
Groups:
- BMS-986165 12 mg BID: Participants receive BMS-986165 12 mg BID for a 12-week double-blind treatment period, then if eligible, move into the 40-week open-label extension period and receive BMS-986165 6 mg BID PO.
- BMS-986165 6 mg BID: Participants were randomized to the 6 mg BID arm under the Original Protocol or Protocol Amendment 01 receive 6 mg BID for the 12-week double-blind treatment period and 6 mg BID in the open-label extension period.
- Placebo BID PO: Participants receive placebo for a 12-week double-blind treatment period, then if eligible, move into the 40-week open-label extension period and receive BMS-986165 6 mg BID PO.
Period: Double-Blind Treatment Period
Arm/Group | BMS-986165 12 mg BID | BMS-986165 6 mg BID | Placebo BID PO
Started (Randomized and Treated) | 26 | 4 | 8
Completed | 19 | 3 | 7
Not Completed | 7 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 1
Not completed — Participant request to discontinue treatment | 1 | 0 | 0
Not completed — Participant withdrew consent | 1 | 1 | 0
Not completed — Other Reasons | 2 | 0 | 0
Period: Open-Label Treatment Period
Arm/Group | BMS-986165 12 mg BID | BMS-986165 6 mg BID | Placebo BID PO
Started | 19 | 3 | 7
Completed | 11 | 0 | 1
Not Completed | 8 | 3 | 6
Not completed — Lack of Efficacy | 0 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 3
Not completed — Participant request to discontinue treatment | 1 | 0 | 0
Not completed — Participant withdrew consent | 1 | 0 | 3
Not completed — Administrative reason by sponsor | 4 | 0 | 0
Not completed — Other reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986165 12 mg BID | BMS-986165 6 mg BID | Placebo BID PO | Total
Number analyzed (Participants) | 26 | 4 | 8 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.8 (14.4) | 28.8 (6.7) | 38.0 (15.1) | 39.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 2 | 2 | 16
  Male | 14 | 2 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 3 | 6 | 33
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 25 | 3 | 7 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Response at Week 12
Description: Clinical response is defined as achieving the following changes in the modified Mayo score (excludes the physicians' global assessment)
  * A decrease from baseline in the modified Mayo score of ≥ 2 points, and
  * A decrease from baseline in the modified Mayo score ≥ 30%, and
  * A decrease in rectal bleeding (RB) subscore of ≥ 1 point or absolute RB subscore ≤ 1
  Note: The modified Mayo score calculated to determine eligibility will also be used as the baseline disease activity score.
  The modified Mayo score is a 9-point scale (a score of 5 to 9 points denotes moderate to severe disease). The modified Mayo score is a sum of the following 3 components:
  * Stool frequency (SF) subscore (0 to 3)
  * Rectal bleeding (RB) subscore (0 to 3)
  * Endoscopic (ES) subscore (0 to 3)
Time Frame: At week 12
Population: Prespecified to be collected for all randomized participants in Arms "BMS-986165 12 mg BID" and "Placebo BID PO". "BMS-986165 6 mg BID" was removed under Protocol Amendment 02.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BMS-986165 12 mg BID | Placebo BID PO
Number analyzed (Participants) | 26 | 8
Percentage of participants | 53.8 [33.4 to 73.4] | 50.0 [15.7 to 84.3]
Statistical Analysis 1: Comparison: BMS-986165 12 mg BID vs Placebo BID PO; Test type: Superiority; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-35.7 to 43.4]

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. Note: the first dose of study treatment in the open-label period may be the same as the last dose date of study treatment in double-blind treatment period, therefore, the participants analyzed in the open-label period may contain double blind participants finishing their last dose in the double-blind treatment period.
Time Frame: From first dose up to the last dose in the double-blind period or 30 days post the last dose date if not treated in the open-label period and from the first dose in open-label period up to 30 days post the last dose date (up to approximately 402 days)
Population: All randomized participants who receive at least 1 dose of double-blind study treatment. Prespecified to be collected for participants in Arms "BMS-986165 12 mg BID" and "Placebo BID PO". "BMS-986165 6 mg BID" was removed under Protocol Amendment 02.
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 12 mg BID | Placebo BID PO
Number analyzed (Participants) | 26 | 8
Participants
  Double-Blind Treatment Period | 21 | 6
  Open-Label Treatment Period | 15 | 6

3. Primary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability or permanent damage, is a congenital anomaly/birth defect, is an important medical event. Note: the first dose of study treatment in the open-label period may be the same as the last dose date of study treatment in double-blind treatment period, therefore, the participants analyzed in the open-label period may contain double blind participants finishing their last dose in the double-blind treatment period.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 12 mg BID | Placebo BID PO
Number analyzed (Participants) | 26 | 8
Participants
  Double-Blind Treatment Period | 4 | 1
  Open-Label Treatment Period | 1 | 1

4. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 12 mg BID | Placebo BID PO
Number analyzed (Participants) | 26 | 8
Participants
  Double-Blind Treatment Period | 2 | 0
  Open-Label Treatment Period | 1 | 3

5. Primary Outcome: Number of Participants Experiencing Adverse Events of Special Interest (AEIs)
Description: An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. AEs of special interest include: skin events, influenza, herpes viral infections, opportunistic infections, tuberculosis, cardiovascular events, malignancy, and COVID-19.
Time Frame: From first dose to 52 weeks after first dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986165 12 mg BID | Placebo BID PO
Number analyzed (Participants) | 26 | 8
Participants
  Skin Events | 15 | 5
  Influenza | 1 | 2
  Herpes Viral Infections | 0 | 0
  Opportunistic Infections | 0 | 0
  Tuberculosis | 0 | 0
  Cardiovascular events | 1 | 0
  Malignancy | 0 | 0
  COVID-19 | 3 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion (up to approximately 420 days). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 402 days)
Groups:
- BMS-986165 12 mg BID (Double-Blind Treatment Period): Participants receive BMS-986165 12 mg BID for a 12-week double-blind treatment period.
- BMS-986165 6 mg BID (Double-Blind Treatment Period): Participants were randomized to the 6 mg BID arm under the Original Protocol or Protocol Amendment 01 receive 6 mg BID for the 12-week double-blind treatment period.
- Placebo BID PO (Double-Blind Treatment Period): Participants receive placebo for a 12-week double-blind treatment period.
- BMS-986165 6 mg BID (Open-Label Treatment Period): Eligible participants that move into the 40-week open-label extension period receive BMS-986165 6 mg BID PO.
Arm/Group | BMS-986165 12 mg BID (Double-Blind Treatment Period) | BMS-986165 6 mg BID (Double-Blind Treatment Period) | Placebo BID PO (Double-Blind Treatment Period) | BMS-986165 6 mg BID (Open-Label Treatment Period)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/4 | 0/8 | 0/29
Serious Adverse Events (participants affected / at risk) | 4/26 | 0/4 | 1/8 | 2/29
Other Adverse Events (participants affected / at risk) | 19/26 | 4/4 | 6/8 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 12 mg BID (Double-Blind Treatment Period) (N=26) | BMS-986165 6 mg BID (Double-Blind Treatment Period) (N=4) | Placebo BID PO (Double-Blind Treatment Period) (N=8) | BMS-986165 6 mg BID (Open-Label Treatment Period) (N=29)
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Bacteroides bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986165 12 mg BID (Double-Blind Treatment Period) (N=26) | BMS-986165 6 mg BID (Double-Blind Treatment Period) (N=4) | Placebo BID PO (Double-Blind Treatment Period) (N=8) | BMS-986165 6 mg BID (Open-Label Treatment Period) (N=29)
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Tongue dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 3 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 8 | 3 | 1 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT04613518/Prot_SAP_000.pdf